CLINICAL TRIAL: NCT06997991
Title: Prospective Clinical Study to Evaluate the Safety and Efficacy of Intraarticular Administration of Micro-grafts of Adipose Tissue (Adipo-micro-grafts) in the Treatment of Osteoarthritis of the Trapezium-metacarpal Joint
Brief Title: Prospective Clinical Study to Evaluate the Safety and Efficacy of Intraarticular Administration of Micro-grafts of Adipose Tissue (Adipo-micro-grafts) in the Treatment of Osteoarthritis of the Trapezium-metacarpal Joint (ADIPO_MICRO_GRAFTS_1)
Acronym: AMG_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Michele Riccio, Director Dpt Reconstructive and Hand Surgery, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1155772|26/07/2022
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis; Osteoarthritis Thumbs
Keywords: adipose stem cells; Rigenera protocol; trapeziometacarpal arthritis; microfragmented adipose tissue
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adipose micro-grafts (Experimental): Patients were positioned supine, and local anesthesia was administered. A small incision was made to introduce a blunt cannula attached to a Luer-lock 60-cc syringe. Klein sterile solution, containing saline and lidocaine, was injected into the subcutaneous fat layer of either the abdominal or thigh region. Subsequently, approximately 30 mL of adipose tissue was extracted. The collected lipoaspirate was processed under sterile conditions in a closed system using Rigenera® technology (HBW, Turin, Italy). Before injecting, the skin was sterilely dressed, and the injection of 2-3 mL of aMAT was performed into TMC joint with a superolateral approach, under fluoroscopic X-ray guidance and using a disposable 20G needle and a 3 mL Luer-Lock Syringe.
  Interventions: Procedure: adipose micro-grafts injection

INTERVENTIONS:
Procedure: adipose micro-grafts injection — Patients were positioned supine, and local anesthesia was administered. A small incision was made to introduce a blunt cannula attached to a Luer-lock 60-cc syringe. Klein sterile solution, containing saline and lidocaine, was injected into the subcutaneous fat layer of either the abdominal or thigh region. Subsequently, approximately 30 mL of adipose tissue was extracted. The collected lipoaspirate was processed under sterile conditions in a closed system using Rigenera® technology (HBW, Turin, Italy). Before injecting, the skin was sterilely dressed, and the injection of 2-3 mL of aMAT was performed into TMC joint with a superolateral approach, under fluoroscopic X-ray guidance and using a disposable 20G needle and a 3 mL Luer-Lock Syringe.

SUMMARY:
The objective of this interventional study is the Change in the Michigan Hand Questionnaire (MHQ) score over time in subjects with Eaton Littler grade II and III trapeziometacarpal osteoarthritis.

The main questions to be answered are:

* primary outcomes: Differences in the change in the MHQ scale measured as a reduction in the score result of 12 points within 6 months from preoperative.
* secondary outcomes: Change from baseline in hand function measured by grip strength (Gripstrength); Change from baseline in hand function by lateral grip strength (tippinch and tripodpinch); Change in the Visual Analogue Scale (VAS) pain scale before the procedure then after the procedure, at 1, 3 and 6 months; Safety and tolerance of the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Male or female aged ≥ 40 and ≤ 75 years
3. Normal axial alignment
4. Eaton/Littler stage 2-3
5. MHQ pain scale
6. Willingness to participate in all scheduled follow-ups
7. Willingness to abstain from taking level 2 analgesics and opioids for the duration of the study. NSAIDs and Paracetamol are permitted.

Exclusion Criteria:

1. Pregnant and/or breastfeeding women.
2. If a woman, of childbearing age and the subject is not using a highly effective method of birth control and is not willing to use it during participation in the clinical trial. Highly effective methods of birth control include: combined hormonal contraception (containing estrogen and progestin) combined with ovulation inhibition (oral, intravaginal, transdermal); progestin-only hormonal contraception combined with ovulation inhibition (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence;
3. Intra-articular injection within 3 months of treatment.
4. Immunocompromised for reasons such as corticosteroid therapy, chemotherapy, antiangiogenic or immunosuppressive agents, or due to immunodeficiency syndromes
5. Previous hand surgery within the last 6 months
6. History of connective tissue disease, such as systemic lupus erythematosus, systemic sclerosis, Sjögren's syndrome or mixed connective tissue disease
7. Infections in the trapezium-metacarpal joint, skin disease or infections in the area of the injection site

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in hand and upper limb function measured by the Michigan Hand questionnaire | The MHQ will be administered at three key time points: before treatment, 3 months, and 6 months after the therapeutic intervention, in order to monitor clinical progress and treatment effectiveness.
  The Michigan Hand Questionnaire (MHQ) is a validated instrument specifically designed to assess hand function and the impact of upper extremity conditions on quality of life. The questionnaire explores six main dimensions: general function, activities of daily living (ADL), pain, aesthetics, patient satisfaction, and work function.
  The score for each domain is converted to a scale of 0 to 100, where:
  100 represents the best perceived functional outcome, 0 represents the worst outcome.
  For some subsections (such as pain), the scale is reversed to ensure correct interpretation of the scores.

SECONDARY OUTCOMES:
Evaluation of: 1. Change from baseline in hand function measured by grip strength 2. Change from baseline in hand function measured by lateral grip strength (tip pinch and tripod pinch) 3. Change in visual analogue scale of pain (VAS) over time 4.Safety | Three key time points: before treatment, 3 months, and 6 months after the therapeutic intervention.
  1. The grip strength of the treated hand is measured with the JAMAR manual hydraulic dynamometer in kilograms of pressure by taking the greatest force of three successive attempts with 15 seconds of rest between each attempt.
  2. The lateral grip strength (tippinch: between the thumb and index finger; tripodpinch: between the thumb, index finger and middle finger) of the treated hand is measured with the mechanical grip meter in kilograms of pressure by taking the greatest force of three successive attempts with 15 seconds of rest between each attempt.
  3. Differences in the pain scale measured as a reduction in pain perception. Pain in the treated joint will be assessed by a visual analogue scale that requires the patient to respond by placing a vertical line on a 100mm scale where 0 corresponds to "no pain" and 100 "unbearable pain".
  4. Evaluation of the safety and tolerability of the treatment, detected by examining the adverse events expected at local level.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Ospedali Riuniti, Ancona, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be shared due to confidentiality and regulatory constraints, except for possible use in scientific publications in anonymized or aggregated format.

REFERENCES:
- [Background] Mayoly A, Witters M, Jouve E, Bec C, Iniesta A, Kachouh N, Veran J, Grimaud F, Zavarro AC, Fernandez R, Bendahan D, Giraudo L, Dumoulin C, Chagnaud C, Casanova D, Sabatier F, Legre R, Jaloux C, Magalon J. Intra Articular Injection of Autologous Microfat and Platelets-Rich Plasma in the Treatment of Wrist Osteoarthritis: A Pilot Study. J Clin Med. 2022 Sep 29;11(19):5786. doi: 10.3390/jcm11195786. PMID 36233654
- [Background] Erne HC, Cerny MK, Ehrl D, Bauer AT, Schmauss V, Moog P, Broer PN, Loew S, Schmauss D. Autologous Fat Injection versus Lundborg Resection Arthroplasty for the Treatment of Trapeziometacarpal Joint Osteoarthritis. Plast Reconstr Surg. 2018 Jan;141(1):119-124. doi: 10.1097/PRS.0000000000003913. PMID 28922320
- [Background] Cook GS, Lalonde DH. MOC-PSSM CME article: Management of thumb carpometacarpal joint arthritis. Plast Reconstr Surg. 2008 Jan;121(1 Suppl):1-9. doi: 10.1097/01.prs.0000294708.70340.8c. PMID 18182958
- [Background] De Francesco F, Gravina P, Busato A, Farinelli L, Soranzo C, Vidal L, Zingaretti N, Zavan B, Sbarbati A, Riccio M, Gigante A. Stem Cells in Autologous Microfragmented Adipose Tissue: Current Perspectives in Osteoarthritis Disease. Int J Mol Sci. 2021 Sep 22;22(19):10197. doi: 10.3390/ijms221910197. PMID 34638538
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Farinelli L, Riccio M, Gigante A, De Francesco F. Pain Management Strategies in Osteoarthritis. Biomedicines. 2024 Apr 4;12(4):805. doi: 10.3390/biomedicines12040805. PMID 38672160